CLINICAL TRIAL: NCT01312805
Title: Using Computers to Assist in the Treatment of Asthma in a Pediatric Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Aaron Carroll, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHICA_Asthma_Study
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: asthma; clinical decision support; CHICA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA Control (Active Comparator): This arm received CHICA without the asthma module
  Interventions: Other: CHICA Control
- CHICA Asthma Module (Experimental): This arm received the CHICA asthma module
  Interventions: Other: CHICA Asthma Module

INTERVENTIONS:
Other: CHICA Asthma Module — This module was added to CHICA to help diagnose and manage asthma
  Arms: CHICA Asthma Module
Other: CHICA Control — This is CHICA without the asthma module, and was used as a control
  Arms: CHICA Control

SUMMARY:
This study seeks to improve physician adherence to four recommendations of the NHLBI asthma treatment guidelines:

1. Improve case detection of asthma among patients with pulmonary symptoms,
2. Grade all asthma patients asthma, identifying those with persistent versus intermittent asthma,
3. Improve rates of use of controller medications - particularly inhaled steroids - among patients with persistent asthma,
4. Provide an asthma treatment plan for all asthma patients.

DETAILED DESCRIPTION:
Objectives: Improve physician adherence to four recommendations of the NHLBI asthma treatment guidelines:

1. Improve case detection of asthma among patients with pulmonary symptoms,
2. Grade all asthma patients asthma, identifying those with persistent versus intermittent asthma,
3. Improve rates of use of controller medications - particularly inhaled steroids - among patients with persistent asthma,
4. Provide an asthma treatment plan for all asthma patients.

Design: This will be a randomized controlled trial. Patients registering for appointments at the PCC Pediatric clinic will be randomized to an intervention or control arm. Patients in the intervention arm, and the physicians who see them, will receive the full intervention. Patients in the control arm will receive usual care.

Intervention: The CHICA computer system has been in regular use at the PCC Pediatrics clinic since November 4, 2004. At patient check-in, CHICA produces a health survey that parents complete in the weighting room. The survey is scanned into CHICA before the physician encounter. CHICA produces a worksheet for the physician that includes prompts and reminders based date from the health survey and the electronic medical record. The completer worksheet is scanned back into CHICA. Intervention and control groups will continue to use this system

In the intervention group, CHICA will include a question asking for the presence of asthma or asthma symptoms on the health survey. If the family responds that asthma or symptoms of asthma are present, CHICA will:

1. Alert the physician and ask him or her to confirm or deny the presence of asthma and to rate the asthma as persistent or intermittent,
2. Generate a chart showing the criteria for each asthma grade,
3. Recommend controller medications if the patient has persistent asthma and ask the physician to document if controllers were prescribed,
4. Generate a partially completed treatment plan for the physician to complete and give to the patient.

For patients confirmed to have asthma, CHICA will place a question on the health survey at subsequent visits that assesses symptoms. For patients who have been prescribed controller medications, CHICA will put a question on the health survey asking about patient adherence to the medication. The physician worksheet will alert the physician to changes in the patient's symptom status or to non-adherence to controller medication, in compliance with NHLBI guidelines.

Outcome Measures: To determine the rates of asthma case finding in the intervention and control groups, we will pull the RMRS electronic records of all patients seen during the first 6 months of the trial and determine the prevalence of diagnoses for asthma (ICD-9 code equal to 493.*).

After 6 months of running the trial, we will randomly select from those patients in the trial who have an ICD-9 diagnosis of asthma (493.*), 75 patients from the intervention group and 75 patients from the control group. The paper "shadow" charts for these patients will be pulled from the chart room at the PCC Pediatrics clinic. Trained chart reviewers will document the following:

1. Has the patient's asthma been graded as intermittent or persistent?
2. Is there documentation of an asthma treatment plan?
3. Has the patient been prescribed a controller medication?

ELIGIBILITY:
Inclusion Criteria:

* Families who visit the Wishard/IUMG Primary Care Center (PCC) pediatric clinic are eligible for our study. Families are randomly assigned to either the control or intervention group, where they will remain for the study's duration. No blocking or other methods of stratification are used. There are no additional exclusion criteria. Data collection will occur for a minimum of 6 months and not to exceed two years

Exclusion Criteria:

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2098 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Wishard Primary Care Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHICA Control | CHICA Asthma Module
Started | 1016 | 1082
Completed | 1016 | 1082
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHICA Control | CHICA Asthma Module | Total
Number analyzed (Participants) | 1016 | 1082 | 2098
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1016 | 1082 | 2098
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 515 | 530 | 1045
  Male | 501 | 552 | 1053

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis Rate of Asthma
Time Frame: one year
Population: We excluded those participants who had a previous diagnosis of asthma in the 14 months before the start of the study. This left the numbers seen above.
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA Control | CHICA Asthma Module
Number analyzed (Participants) | 937 | 1010
Participants | 54 | 87

ADVERSE EVENTS:
Arm/Group | CHICA Control | CHICA Asthma Module
Serious Adverse Events (participants affected / at risk) | 0/1016 | 0/1082
Other Adverse Events (participants affected / at risk) | 0/1016 | 0/1082

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No